CLINICAL TRIAL: NCT07240467
Title: Safety and Efficacy of Bovis Calculus Stativus in the Treatment of Acute Cerebral Ischemic Stroke With Impaired Consciousness- A Multicenter, Prospective, Double-blind, Randomized Trial
Brief Title: Bovis Calculus Stativus Treat Acute Cerebral Ischemic Stroke With Impaired Consciousness
Acronym: ASCENT-BC
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xiang Luo (Other)
Collaborators: The Fifth Hospital of Wuhan (Other); Jingzhou Hospital of Traditional Chinese Medicine (Unknown); Xiangyang Hospital of Traditional Chinese Medicine (Unknown); Wuhan Hospital of Traditional Chinese Medicine (Other); Hubei Hospital of Traditional Chinese Medicine (Other); Wuhan No.1 Hospital (Other); Wuhan Central Hospital (Other); Xiangyang No.1 People's Hospital (Other); Taihe Hospital affiliated to Hubei University of Medicine (Unknown); Yichang Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Xiang Luo, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20250712
Record Dates: First submitted 2025-11-16; First posted 2025-11-21 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke AIS; Impaired Consciousness
Keywords: acute ischemic stroke; impaired consciousness; Bovis Calculus Stativus
MeSH Terms: conditions — Ischemic Stroke | interventions — Long-Term Synaptic Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bovis Calculus Stativus (BCS) group (Experimental): Patients with acute ischemic stroke accompanied by impaired consciousness within 72 hours and a Glasgow Coma Scale (GCS) score of 3-12, who are randomized to the experimental group, will be administered 0.6 g of BCS orally or via nasogastric tube immediately after recruitment. Subsequently, in accordance with guidelines, they will receive standard acute stroke treatment along with 0.6 g of BCS twice daily (bid) orally or via nasogastric tube for 5 consecutive days.
  Interventions: Drug: Bovis Calculus Stativus (BCS)
- placebo group (Placebo Comparator): Patients with acute ischemic stroke accompanied by impaired consciousness within 72 hours and a GCS score of 3-12, who are randomized to the control group, will be administered a placebo following the same regimen after recruitment. Subsequently, in accordance with guidelines, they will receive standard acute stroke treatment along with the placebo administered orally or via nasogastric tube for 5 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bovis Calculus Stativus (BCS) — Patients with acute ischemic stroke accompanied by impaired consciousness within 72 hours and a Glasgow Coma Scale (GCS) score of 3-12, who are randomized to the experimental group, will be administered 0.6 g of BCS orally or via nasogastric tube immediately in the emergency room. Subsequently, in accordance with guidelines, they will receive standard acute stroke treatment along with 0.6 g of BCS twice daily (bid) orally or via nasogastric tube for 5 consecutive days.
  Other Names: trade: Bovis Calculus Stativus (BCS);Wuhan Jianmin Dapeng Pharmaceutical Co., Ltd.
  Arms: Bovis Calculus Stativus (BCS) group
Drug: Placebo — Patients with acute ischemic stroke accompanied by impaired consciousness within 72 hours and a GCS score of 3-12, who are randomized to the control group, will be administered a placebo following the same regimen in the emergency room. Subsequently, in accordance with guidelines, they will receive standard acute stroke treatment along with the placebo administered orally or via nasogastric tube for 5 consecutive days.
  Arms: placebo group

SUMMARY:
Acute ischemic stroke (AIS) is a severe and life-threatening condition, with 35% of AIS patients experiencing impaired consciousness upon admission within 24 hours of onset. Previous studies indicated that patients with impaired consciousness at the onset of stroke have a higher incidence of stroke-related complications, particularly cerebral edema and pneumonia, as well as higher in-hospital and three-month mortality rates. The etiology of impaired consciousness in AIS is complex: ischemic damage to reticular activating system of the brainstem can directly lead to cell necrosis and result in impaired consciousness. Furthermore, secondary pathological changes following AIS, such as excitatory amino acid toxicity, oxidative stress, free radical production, and cascading inflammatory responses, can indirectly worsen impaired consciousness. Therefore, impaired consciousness at the onset of AIS is the result of cellular damage under multiple pathophysiological mechanisms. Developing neuroprotective drugs with multiple targets is key to effectively improving adverse outcomes related to impaired consciousness in AIS. However, there is currently a lack of treatment specifically aimed at improving impaired consciousness at the onset of AIS.

Cultivated Bovine Bezoar (Bovis Calculus Stativus, BCS) combines the advantages of pharmacological similarity to natural bovine by adding components such as deoxycholic acid, cholic acid, and composite calcium bilirubin to fresh bovine bile. It is rich in various trace elements and amino acids and is a compound medication that can exert neuroprotective effects through multiple pathways and targets. In traditional Chinese medicine, it has long been used to treat various consciousness disorder-related diseases, including stroke. The various components of in vitro cultivated bezoar are also widely used in clinical research for various neurological diseases.The above evidence fully demonstrates that BCS is an optimal treatment for impaired consciousness in stroke.

The goal of this clinical trial is to learn if Bovis Calculus Stativus works to treat acute cerebral ischemic stroke with impaired consciousness. It will also learn about the safety of Bovis Calculus Stativus. The main questions it aims to answer are:

1. Does Bovis Calculus Stativus treat and alleviate consciousness disorders in patients with acute cerebral infarction accompanied by impaired consciousness ？
2. What medical problems do participants have when taking Bovis Calculus Stativus?

Researchers will compare Bovis Calculus Stativus to a placebo (a look-alike substance that contains no drug) to see if Bovis Calculus Stativus works to treat acute cerebral ischemic stroke with impaired consciousness.

Participants will:

1. receive treatment with Bovis Calculus Stativus (or placebo) for 5 days.
2. Take an in-person or telephone follow-up within 90 days after the acute stroke.

DETAILED DESCRIPTION:
This study evaluates whether the combination of Bovis Calculus Stativus (BCS) with conventional treatment can improve impaired consciousness and functional outcomes, and whether it increases serious adverse events in patients with acute cerebral infarction accompanied by impaired consciousness within 72 hours of onset. This is a prospective multicenter randomized controlled double-blind study. In 12 centers in China,220 patients with the following situations will be enrolled: acute ischemic stroke accompanied by impaired consciousness within 72 hours and a GCS score of 3-12. Patients will be randomly assigned into 2 groups according to the ratio of 1:1:

1. Experimental Group:

   Patients with acute ischemic stroke accompanied by impaired consciousness within 72 hours and a Glasgow Coma Scale (GCS) score of 3-12, who are randomized to the experimental group, will be administered 0.6 g of BCS orally or via nasogastric tube immediately after recruitment. Subsequently, in accordance with guidelines, they will receive standard acute stroke treatment along with 0.6 g of BCS twice daily (bid) orally or via nasogastric tube for 5 consecutive days.
2. Placebo Control Group:

Patients with acute ischemic stroke accompanied by impaired consciousness within 72 hours and a GCS score of 3-12, who are randomized to the control group, will be administered a placebo following the same regimen immediately after recruitment. Subsequently, in accordance with guidelines, they will receive standard acute stroke treatment along with the placebo administered orally or via nasogastric tube for 5 consecutive days.

Patients will be assessed using the GCS and NIHSS scores at 24 hours and 8 days after randomization, and the mRS score at 8 days after randomization. A follow-up visit, either in person or via telephone, will be conducted 90 days after randomization to assess the mRS and EQ-5D-5L scores.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Clinically diagnosed with ischemic cerebral infarction;
* GCS score: 3-12;
* Time from symptom onset to randomization ≤ 24 hours, including wake-up stroke or stroke without a witness; the time of symptom onset is defined as the "last known well time";
* Pre-stroke mRS score of 0-1;
* Head CT excludes intracranial hemorrhage or other non-ischemic pathologies;
* The participant or legally authorized representative is capable of providing informed consent.

Exclusion Criteria:

* Use of in BCS within 24 hours before treatment;
* Known pregnancy or breastfeeding, or positive pregnancy test before randomization;
* Allergy to BCS;
* Impaired consciousness caused by other diseases, such as metabolic disorders (e.g., ketoacidosis), trauma, infectious diseases (e.g., pneumonia), neoplastic diseases (e.g., glioma), or toxic conditions (e.g., organophosphate poisoning);
* Requiring or undergoing hemodialysis or peritoneal dialysis; known severe renal insufficiency (glomerular filtration rate <30 mL/min or serum creatinine >220 μmol/L);
* Expected survival time less than 6 months (e.g., due to malignancy, severe cardiopulmonary disease, etc.);
* Participation in other interventional clinical studies that may affect outcome assessment;
* Other conditions deemed by the investigator to make the patient unsuitable for participation or pose significant risks (e.g., inability to understand and/or comply with study procedures and/or follow-up due to mental illness, cognitive or emotional disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2028-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with GCS improvement ≥2 points | Day 8 after randomization
  Proportion of patients with a GCS score increase of 2 points or more to assess the improvement rate of impaired consciousness

SECONDARY OUTCOMES:
GCS shift analysis | Day 8 after randomization
  GCS score overall shift assessment of consciousness disturbance overall improvement ratio
Proportion of mRS 0-2 | Day 90 after randomization
  Proportion of overall favorable prognosis
Proportion of NIHSS score 0-1 or a reduction of ≥4 points from baseline | Day 8 after randomization
  Proportion of good neurological function recovery
EQ-5D-5L index score | Day 90 after randomization
  The EQ-5D-5L index score is a single summary number that represents a person's overall health state based on the EQ-5D-5L descriptive system. It's a crucial tool for calculating Quality-Adjusted Life Years (QALYs) used in health economics and outcomes research.The five levels are:
  * Level 1: No problems
  * Level 2: Slight problems
  * Level 3: Moderate problems
  * Level 4: Severe problems
  * Level 5: Extreme problems / Unable to
In-hospital stroke-associated pneumonia incidence rate | Day 8 after randomization
  Proportion of Hospital-Acquired Pneumonia Complications

OTHER OUTCOMES:
The incidence of SAE | Day 8 after randomization
  The incidence of SAE
All-cause mortality | Day 8 after randomization
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Xiang Luo, PhD MD, Principal Investigator — Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei 450001; Xiang Luo, PhD MD, Principal Investigator — Tongji Hospital Affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guo Y, Yan S, Xu L, Zhu G, Yu X, Tong X. Use of angong niuhuang in treating central nervous system diseases and related research. Evid Based Complement Alternat Med. 2014;2014:346918. doi: 10.1155/2014/346918. Epub 2014 Dec 18. PMID 25587341